CLINICAL TRIAL: NCT07388277
Title: A Phase I/II Study of CC-97540 (BMS-986353), CD19-Targeted NEX-T CAR T Cells, in Patients With Antineutrophil Cytoplasmic Antibody-associated Vasculitis
Brief Title: CC-97540 in Patients With Antineutrophil Cytoplasmic Antibody-associated Vasculitis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Marcela V. Maus, M.D.,Ph.D. (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Marcela V. Maus, M.D.,Ph.D., Sponsor-Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P003179
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Antineutrophil Cytoplasmic Antibody-associated Vasculitis
Keywords: Refractory/Relapsing ANCA-associated vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-97540 (Experimental): Prior to receiving CC-97540, participants will undergo lymphodepleting chemotherapy. Lymphodepleting chemotherapy is the combination of cyclophosphamide and fludarabine and will be administered intravenously. CC-97540 will be infused intravenously on day 0 only.
  Interventions: Drug: CC-97540; Drug: Lymphodepletion Chemotherapy

INTERVENTIONS:
Drug: CC-97540 — Intravenous infusion
  Other Names: BMS-986353; CD19-Targeted NEX-T CAR T Cells
Drug: Lymphodepletion Chemotherapy — Intravenous infusion of cyclophosphamide and fludarabine

SUMMARY:
The purpose of this study is to evaluate the safety of CC-97540 in relapsed or refractory severe antineutrophil cytoplasmic antibody (ANCA)-associated vasculitis.

DETAILED DESCRIPTION:
This is a two-part, non-randomized, open label, single site Phase I/II study to assess the safety and efficacy of CC-97540 CAR T cell products for treatment of relapsing or refractory ANCA-associated vasculitis. This study consists of 2 parts: Part A (Safety Lead-In), a verification of the safety of the infusion dose, and Part B (Expansion), in which participants receive CC-97540 CAR T cells at the dose confirmed in Part A.

This is a Phase I/II clinical trial. Phase I/II clinical trials test the safety and effectiveness of an investigational therapy to learn whether the therapy works in treating a specific disease. "Investigational" means that the therapy is being studied.

The U.S. Food and Drug Administration (FDA) has not approved CC-97540 as a treatment for any disease.

It is expected that about 12 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Able to voluntarily provide written informed consent prior to the performance of any study-specific procedures.

  -≥18 years of age at the time of signing informed consent.
* Classification as granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA) per the American College of Rheumatology (ACR) / European Alliance of Associations for Rheumatology (EULAR) 2022 definitions (Robson et al., 2022, Suppiah et al., 2022) (see Appendix A).
* Current or historical positive proteinase 3 (PR3) or myeloperoxidase (MPO) antibody testing or a cytoplasmic (cANCA) or perinuclear antineutrophil cytoplasmic antibody (pANCA) immunofluorescence pattern. (Antibodies and immunofluorescence may currently be negative.)
* Active ANCA-associated vasculitis within 6 weeks of screening presenting as either:
* Relapsed disease (BVASv3 > 0 following prior remission) despite standard-of-care treatment per the ACR/Vasculitis Foundation (VF) Guidelines for the Management of ANCA-Associated Vasculitis (Chung et al., 2021), or
* Refractory disease (persistent BVASv3 positivity) despite standard-of-care treatment per the ACR/VF Guidelines (Chung et al., 2021). Refractory disease is defined as persistent BVASv3 positivity despite at least 6 weeks of appropriate guideline-indicated standard-of-care treatment per the ACR/VF Guidelines for the Management of ANCA-Associated Vasculitis.

Appropriate guideline-indicated standard-of-care treatment per the ACR/VF Guidelines for the Management of ANCA-Associated Vasculitis includes:

* either rituximab or cyclophosphamide for severe disease;
* or, methotrexate or azathioprine for non-severe disease.

  -Severe disease activity defined as:
* 1 or more major BVAS/WG criteria or at least 3 minor BVASv3 items (see Appendix B), or
* 1 or more of cutaneous ulceration, retroorbital disease, sinonasal disease with bony or cartilage damage, subglottic stenosis, or renal involvement, or
* Unanimous expert committee consensus on severity (3/3 agreement).

  * Left ventricular ejection fraction > 45%.
  * Adequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) <2.5 × upper limit of normal (ULN) and direct bilirubin <1.5 × ULN. Elevation in bilirubin attributable to Gilbert's syndrome is permitted.
  * Adequate renal function defined by creatinine clearance >30 ml/min using the Cockcroft-Gault formula. Measured creatinine clearance from a 24-hour urine collection is acceptable if clinically indicated. For select subjects, including those with short stature or low lean muscle mass, alternative calculators to Cockcroft-Gault such as Modification in Diet Renal Disease (MDRD), Chronic Kidney Disease Epidemiology (CKD-EPI), or Cystatin C measurements may be used.
  * Absolute lymphocyte count of ≥ 300 cells/uL.
  * Adequate organ function defined as:
* Hemoglobin ≥ 8 g/dL
* Platelet count ≥ 75,000/uL

  * Willingness to adhere to contraceptive requirements. The effects of CC-97540 CAR T cells on the developing human fetus are unknown. Lymphodepleting chemotherapy poses genotoxic, fetotoxic, and infertility risks. For these reasons, women of child-bearing potential and men with partners of childbearing potential must use effective contraception beginning prior to leukapheresis and continuing for at least 12 months after CC-97540 infusion. Due to potential unknown interactions of CC-97540 with hormonal contraception, an additional barrier method should be used if hormonal contraception is chosen. Participants who become pregnant or suspect pregnancy during the study must notify the treating physician immediately.
  * Ability and willingness to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

* Current or historical positivity for a glomerular basement membrane antibody.
* ANCA-associated vasculitis deemed drug-induced or cocaine/levamisole-associated.
* Treatment of relapsing disease with rituximab or other B cell-depleting therapy for the current episode of relapsed vasculitis. Prior rituximab use for a prior episode (flare) of vasculitis activity is permitted.
* Parkinson's disease, epilepsy, aphasia, cerebellar disease.
* Prior organ transplant currently requiring an immunosuppressive regimen.
* Active malignancy requiring treatment other than non-metastatic basal cell or squamous cell skin carcinoma.
* Treatment with any prior CAR T cell therapy.
* Significant comorbid condition or disease which in the judgment of the Principal Investigator would place the subject at undue risk or interfere with the study.
* Active, uncontrolled, systemic bacterial, viral, or fungal infection.
* Subjects with a history of class III or IV congestive heart failure or with a history of non- ischemic cardiomyopathy.
* Subjects with unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the previous 3 months.
* Subjects with high bleeding risk including INR or PTT greater than 1.5 times the upper limit of normal unless due to a stable dose of anticoagulation. Ongoing anticoagulation permitted if a stable regimen.
* Absolute neutrophil count < 500 cells/uL.
* Symptomatic cerebrovascular disease or peripheral vascular arterial disease requiring ongoing therapeutic anticoagulation or dual antiplatelet therapy or other vascular disease not allowing for holding of DAPT.
* Subjects with a history of pulmonary embolism (PE) or deep vein thrombosis (DVT) within 6 months of beginning lymphodepletion requiring ongoing anticoagulation.
* Pregnant or lactating women. Pregnant women are excluded from this study because CC-97540 CAR T cell drug products are agents with the potential for adverse effects for a fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CC-97540 T cell drug products, breastfeeding should be discontinued if the mother is treated with CC-97540 CAR T cell drug product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-07-09 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of CC-97540 in ANCA-Associated Vasculitis | Study drug infusion (day 0) to 28 days post study drug infusion, assessed up to 12 months post study drug infusion.
  The occurrence of DLT is the primary endpoint and will be assessed for all patients treated at the expansion dose.
Efficacy of CC-97540 | Study drug infusion (day 0) to 28 days post study drug infusion, assessed up to 12 months post study drug infusion.
  This will be determined by the percentage of participants in treatment-free remission defined as a BVASv3 of 0 off immunosuppressive therapy.

SECONDARY OUTCOMES:
Number of Adverse Events | Study drug infusion (day 0) to 28 days post study drug infusion, assessed up to 12 months post study drug infusion.
  Adverse events will be classified and graded according to the CTCAE v.5.0. This will be determined by the proportion of participants experiencing treatment-related serious AEs.
6 Months Treatment-Free Remission | Study drug infusion (day 0) to 28 days post study drug infusion, assessed up to 6-months following study drug infusion.
  Determined by the percentage of participants in treatment-free remission.
6 Months Sustained Treatment-Free Remission | Study drug infusion (day 0) to 28 days post study drug infusion, assessed up to 6-months following study drug infusion.
  Determined by the percentage of participants in sustained treatment-free remission BVASv3 of 0 without use of immunosuppressive therapy since CAR T cell infusion.
12 Months Sustained Treatment-Free Remission | Study drug infusion (day 0) to 28 days post study drug infusion, assessed up to 12 months post study drug infusion.
  Determined by the percentage of participants in sustained treatment-free remission at 12 months following infusion of CC-97540.
Severe and Non-Severe ANCA-Associated Vasculitis | Study drug infusion (day 0) to 28 days post study drug infusion, assessed up to 12 months post study drug infusion.
  Determined by the percentage of participants with severe and non-severe ANCA-associated vasculitis relapse by 6 and 12 months following infusion of CC-97540 with severe relapse defined as 1 or more new or worsened major BVASv3 item or 3 or more minor BVASv3 items and non-severe relapse as 1 or 2 new or worsened minor BVASv3 items.
Time to Severe or Non-Severe Relapse | Study drug infusion (day 0) to 28 days post study drug infusion, assessed up to 12 months post study drug infusion.
  Determined by the time to severe or non-severe relapse following infusion of CC-97540.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Unizony, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation